CLINICAL TRIAL: NCT06356077
Title: SHINE Study: Blood Pressure Evolution and User Satisfaction in a Hypertensive Population Using the Aktiia 24/7 Optical Blood Pressure Monitoring (OBPM) Device: a Prospective Observational Cohort Study.
Brief Title: SHINE: Trends and Satisfaction in Hypertensives Using Aktiia Optical BP Monitoring Device (SHINE)
Acronym: SHINE
Status: Completed | Type: Observational
Sponsor: Aktiia SA (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Other Study IDs: SHINE
Record Dates: First submitted 2024-03-20; First posted 2024-04-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study cohort: Each study subject will receive an Aktiia device and will use it continuously for 3 months. Study participants will have to complete 2 different surveys: one at baseline, and one after the 3 months of Aktiia device use to give their perception on the Aktiia device use as compared to other blood pressure monitors currently on the market.

SUMMARY:
The SHINE study aims to gather data on the evolution of participant's blood pressure and to correlate this with demographic, lifestyle and health factors in a hypertensive population as well as, to gather data on participants' perception of the device under test (Aktiia 24/7).

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants aged 22 to 85 years old
2. A participant whose last blood pressure reading was within the last 12 months and was either:

   1. SBP ≥145
   2. or ≥DBP 90
3. People who use either an iOS or Android smartphone
4. People who have 2 arms
5. Able and willing to provide informed consent and to adhere to study procedures.

Exclusion Criteria:

1. Participants whose BP data submitted is >180 mm Hg systolic OR >120 mm Hg diastolic .
2. Participants with a self-reported known diagnosis of

   1. atrial fibrillation
   2. congestive heart failure
   3. heart valve disease
   4. pheochromocytoma
   5. Raynaud's disease
   6. arm lymphedema
3. Participants who take insulin
4. Participants who are on hemodialysis
5. Women who are self-reported to be pregnant
6. Participants whose arms shake uncontrollably or are paralyzed (cannot move)
7. Participants with upper arm circumference <22 cm or >42 cm
8. Participants with wrist circumference >23cm
9. Participation in another interventional clinical study or use of investigational drugs in the last 30 days.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The final study population should cover the following phenotypes:
  * Close to 50% females and 50% males,
  * At least 20% of non-Caucasian participants,
  * At least 20% of participants with Systolic Blood Pressure (SBP) ≥150mmHg (assessed at baseline via the study device).
Sampling Method: Non-Probability Sample
Enrollment: 1729 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Blood Pressure evolution over 12 weeks | 3 months
  Means, medians, standard deviations, and ranges for Blood Pressure readings and changes in Blood Pressure readings within the study population between week 1 to week 12.

SECONDARY OUTCOMES:
Preferences of subjects regarding the method to monitor their blood pressure between Aktiia Bracelet, Home Blood Pressure Monitor, or Ambulatory Blood Pressure Monitor | 3 months
  Number of participants with preferences using Aktiia 24/7 device, as copared to Home Blood Pressure Monitor, or Ambulatory Blood Pressure Monitor to monitor their blood pressure.
Correlation between the data from Aktiia 24/7 device continual BP monitoring with sociodemographic, lifestyle and health factors. | 3 months
  Statistics on a potential correlation between Blood Pressure measurements and subjects responses to questionnaires regarding their lifestyle, socioeconomic environment and general health.

CONTACTS AND LOCATIONS:
Locations (1):
- Lindus Health, London, United Kingdom